CLINICAL TRIAL: NCT00972933
Title: Neoadjuvant Anti-CTLA4 Blockade With Ipilimumab in Patients With AJCC Stage IIIB-C (Tx,1-4, N1b,2b, 2c, 3, M0) Melanoma: Immunogenicity And Biomarker Analysis
Brief Title: Immunogenicity and Biomarker Analysis of Neoadjuvant Ipilimumab for Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-144
Record Dates: First submitted 2009-09-03; First posted 2009-09-09 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Melanoma
Keywords: Immunogenicity Analysis; Biomarker Analysis; experimental
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab (Experimental): Induction ipilimumab 10 mg/kg IV day 0, 21 (baseline, week 3) Maintenance Ipilimumab 10 mg/kg IV days 63 (+28 days) and, 84 (+28 days) - (3 weeks apart, starting 2-4 weeks following definitive lymphadenectomy)
  Interventions: Drug: ipilimumab

INTERVENTIONS:
Drug: ipilimumab — Excisional Biopsy - baseline Induction ipilimumab 10 mg/kg IV day 0, 21 - baseline and week 3 Complete lymph node dissection - week ≥ 6 Maintenance Ipilimumab 10 mg/kg IV - Days 63 (+28 days) and, 84 (+28 days) - (3 weeks apart, starting 2-4 weeks following definitive lymphadenectomy)
  Other Names: MDX-010; Yervoy; BMS-734016

SUMMARY:
Ipilimumab is a manufactured monoclonal antibody, much like the antibodies usually made by the human body to fight off infection; however it is not known why the human body does not "fight off" a cancerous tumor. The idea behind developing this experimental drug is to stimulate the immune system to make antibodies to kill cancer cells. This research study is considered "experimental" because it has not received approval from the Food and Drug Administration (FDA) for the treatment of this type of cancer.

This monoclonal antibody has been specifically made to block Cytotoxic T Lymphocyte Antigen 4 (CTLA4), which is a protein found on cells of the immune system. CTLA4 seems to slow down the immune response, so blocking it with an anti-CTLA4 antibody may make the immune response more active. The purpose of this study is to see if Ipilimumab affects the response of the patient's immune system toward their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histologic diagnosis of melanoma belonging to T1-4 N1b,2b,2c,3 M 0 AJCC stages, that may present as any of the following groups:
* Primary melanoma with clinically apparent (overt) regional lymph node metastases, confirmed by pathological diagnosis (biopsy).
* Clinically detected recurrence of melanoma at the proximal regional lymph node(s) basin, confirmed by pathological diagnosis (biopsy).
* Clinically or histologically detected primary melanoma involving multiple regional nodal groups, confirmed by pathological diagnosis (biopsy).
* Clinically detected single site of nodal metastatic melanoma arising from an unknown primary, confirmed by pathological diagnosis (biopsy).
* Patients are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal metastasis, or at the time of clinically detected nodal recurrence. Patients must undergo biopsy (punch) or open biopsy (if done as part of a clinically indicated baseline diagnostic procedure) within 14 days of entry into the study. Lymphadenectomy will be performed after at least 2 and generally not longer than 4 weeks of ipilimumab therapy. Additional delays for definitive lymphadenectomy are allowed if clinically indicated while awaiting the resolution of potential adverse events from ipilimumab therapy.
* Patients must have been evaluated by standard-of-care full body imaging studies (CT, PET-CT or MRI) as part of the initial clinical work-up at baseline (no more than 4 weeks prior to study enrollment) and after completion of 2 doses of ipilimumab (at 6-8 weeks after the first dose of ipilimumab and prior the definitive lymphadenectomy procedure).
* Required values for initial laboratory tests:

  * White Blood Cell ≥ 3000/uL
  * Absolute Neutrophil Count ≥ 1500/uL
  * Platelets ≥ 100 x 103/uL
  * Hemoglobin ≥ 10 g/dL
  * Creatinine ≤ ULN
  * AST/ALT ≤ 2.5 x Upper Limit of Normal (ULN)
  * Bilirubin ≤ ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
  * PT/PTT ≤ ULN (No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.)
* Adequate performance status (ECOG 0, 1).
* Men and women, ≥ 18 years of age.
* Women of childbearing potential (WOCBP) must be willing to use an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of ipilimumab. WOCBP include any female who has experienced menarche and who has not undergone a successful surgical sterilization procedure (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

  * Amenorrhea ≥ 12 consecutive months without another cause, or
  * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.
* Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.

Exclusion Criteria:

* Patients with clinical, radiological/laboratory, or pathological evidence of distant metastatic disease.
* Patients with evidence of soft tissue involvement by gross extranodal extension of tumor manifest by fixation to the fascia, or matting of nodal tissue that would compromise surgical resection as determined by the surgical oncologist.
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Patients with underlying heart conditions who are deemed ineligible for surgery by cardiology consult.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA-4 inhibitor or agonist.
* A history of prior radiotherapy, chemotherapy, including infusion or perfusion therapy for his current disease or any immunotherapy including tumor vaccines, interferon-alfa, interleukins, levamisole or other biologic response modifiers within the past 4 weeks.
* Concomitant therapy with any of the following: IL 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids; unless discontinued ≥ 4 weeks.
* Women of childbearing potential (WOCBP), defined above in Section 4.1, who:
* are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
* have a positive pregnancy test at baseline, or
* are pregnant or breastfeeding.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.

Before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test before first receiving ipilimumab. If the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07-17 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
To study the effects of ipilimumab upon the host immune response in nodal metastatic melanoma and in the peripheral blood comparing pre-treatment with post-treatment (baseline, 6 weeks) immunologic features. | 2.5 years

SECONDARY OUTCOMES:
To study the effects of ipilimumab upon the host immune response. | 2.5 years
To collect pilot data comparing pre-treatment with post-treatment proteomic and genetic features. | 2 years
To evaluate the clinical efficacy of preoperative neoadjuvant therapy with ipilimumab in high risk clinically and pathologically node-positive melanoma patients (AJCC stage IIIB-C). | 5 years
To collect safety data and evaluate the safety of neoadjuvant therapy with ipilimumab in high risk clinically and pathologically node-positive melanoma patients (AJCC stage IIIB-C). | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — UPMC/UPCI
Locations (1):
- University of Pittsburgh Medical Center/University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kobeissi I, Eljilany I, Achkar T, LaFramboise WA, Santana-Santos L, Tarhini AA. A Tumor and Immune-Related Micro-RNA Signature Predicts Relapse-Free Survival of Melanoma Patients Treated with Ipilimumab. Int J Mol Sci. 2023 May 3;24(9):8167. doi: 10.3390/ijms24098167. PMID 37175874
- [Derived] Retseck J, Nasr A, Lin Y, Lin H, Mendiratta P, Butterfield LH, Tarhini AA. Long term impact of CTLA4 blockade immunotherapy on regulatory and effector immune responses in patients with melanoma. J Transl Med. 2018 Jul 4;16(1):184. doi: 10.1186/s12967-018-1563-y. PMID 29973204
- [Derived] Tarhini AA, Zahoor H, Lin Y, Malhotra U, Sander C, Butterfield LH, Kirkwood JM. Baseline circulating IL-17 predicts toxicity while TGF-beta1 and IL-10 are prognostic of relapse in ipilimumab neoadjuvant therapy of melanoma. J Immunother Cancer. 2015 Sep 15;3:39. doi: 10.1186/s40425-015-0081-1. eCollection 2015. PMID 26380086